CLINICAL TRIAL: NCT04241861
Title: Physiological Comparison of High-flow Nasal Cannula, Helmet Pressure Support Ventilation and Continuous Positive Airway Pressure During Acute Hypoxemic Respiratory Failure: a Randomized Cross-over Study
Brief Title: High-flow Nasal Cannula vs. Helmet PSV vs. Helmet CPAP During Respiratory Failure
Acronym: HIGHFLOWHELMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2693
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-01

CONDITIONS: Respiratory Failure; Hypoxemia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-flow oxygen therapy (Experimental): Nasal high flow oxygen therapy will be delivered with the Optiflow system. Initial set flow will be ≥ 50 /min and flows will be decreased in case of intolerance and/or according to patients' requirements: flows≥30 L/min will be mandatory in all enrolled patients. Humidification chamber (MR860, Fisher and Paykel healthcare, New Zealand) will be set at 37 °C or 34 °C according to patient's comfort33. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%.
  Interventions: Other: Respiratory support (High-flow oxygen therapy)
- Helmet PSV (Experimental): Dedicated helmets for noninvasive ventilation will be used and size will be chosen according to neck circumference or according to manufacturer recommendations.
  Each patient will be connected to a compressed-gas based ventilator through a bitube circuit with no humidification.
  The ventilator will be set in PSV, with the following suggested settings 34-38:
  1. initial pressure support≥8-10 cmH2O and adequate to permit of a peak in the inspiratory flow of 100 l/min;
  2. positive end-expiratory pressure=10-12 cmH2O and increased to achieve the oxygenation target according to the choice of the attending physician.
  3. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%.
  4. Inspiratory flow trigger = 1 l/min or according to the practice of each institution;
  5. fastest pressurization time;
  6. expiratory trigger: 10-50% of the maximum inspiratory flow;
  7. maximum inspiratory time 1.2 second.
  Interventions: Other: Respiratory support (Helmet PSV)
- Helmet CPAP (Experimental): Dedicated helmets for noninvasive ventilation will be uses and size will be chosen according to neck circumference or according to manufacturer recommendations.
  Treatment will be delivered through a high-flow generator. The following settings will be applied:
  1. Continuous air flow=50-60 L/min.
  2. Expiratory positive end-expiratory pressure valve set to achieve a PEEP==10-12 cmH2O and eventually increased to achieve the oxygenation target according to the choice of the attending physician.
  3. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%. Pressure inside the helmet will be monitored with a manometer in order to maintain the set PEEP.
  Interventions: Other: Respiratory support (Helmet CPAP)

INTERVENTIONS:
Other: Respiratory support (High-flow oxygen therapy) — Noninvasive respiratory support respiratory support
  Arms: High-flow oxygen therapy
Other: Respiratory support (Helmet PSV) — Noninvasive respiratory support respiratory support
  Arms: Helmet PSV
Other: Respiratory support (Helmet CPAP) — Noninvasive respiratory support respiratory support
  Arms: Helmet CPAP

SUMMARY:
The investigators designed a cross-over, randomized trial to assess the physiological effects of helmet pressure support ventilation (PSV) and continuous positive airway pressure (CPAP) as compared to high-flow nasal cannula during the early phase of acute hypoxemic respiratory failure

DETAILED DESCRIPTION:
Setting: 21-bed general ICU, emergency room of the Emergency department (ED), Fondazione Policlinico Universitario "Agostino Gemelli" IRCCS, Rome, Italy..

Patients: adult hypoxemic non-hypercapnic patients admitted to the emergency department or the ICU with de novo acute respiratory failure will be assessed for the enrolment.

Each eligible patient, in the absence of exclusion criteria, will receive 15 minutes of heated and humidified 60% oxygen at a rate of 50 l/min via a non-rebreathing face mask. An ABG will be then collected and PaO2/FiO2 ratio computed: given the high flows used, actual FiO2 will be approximated to the set one.

Nonhypercapnic patients with a PaO2/FiO2≤200 mmHg will be enrolled. In the absence of exclusion criteria and if all other inclusion in criteria are met, patients showing PaO2/FiO2≤300 and >200 mmHg will be treated according to the clinical practice eventually reassessed for the presence of oxygenation criterion subsequently.

Enrolled patients will receive all the interventions (helmet CPAP, PSV and high-flow nasal cannula) in a randomized, cross-over fashion, for 40 minutes each.

At the end of the study, the patient will receive the treatment that will be shown as more appropriate for the patient, according to the attending physician, who will be informed about the results of the study on the individual patient.

ELIGIBILITY:
Inclusion Criteria:

Patients: adult hypoxemic non-hypercapnic patients admitted to the emergency department or the ICU with de novo acute respiratory failure will be assessed for the enrolment.

Patients will be considered eligible whether all the following inclusion criteria are met:

1. Respiratory rate>25 bpm.
2. PaO2/FiO2 ≤200 in the supine position, measured after 15 minutes of high flow treatment with face mask (60 l/min, temperature of the humidification chamber set at 37°C, FiO2 set to achieve a SpO2 >92% and <98%). Given the use of the high flows, nominal FiO2 will be considered a reliable estimate of the actual one.
3. PaCO2 <45mmHg
4. Absence of history of chronic respiratory failure or moderate to severe cardiac insufficiency.
5. Written informed consent

Exclusion Criteria:

* Exacerbation of asthma or chronic obstructive pulmonary disease;
* Cardiogenic pulmonary oedema;
* Haemodynamic instability (Systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg) and/or lactic acidosis (lactate >5 mmol/L) and/or clinically diagnosed Shock
* Metabolic Acidosis (pH <7.30 with normal- or hypo-carbia);
* Glasgow coma scale <13;
* Recent head surgery or anatomy that prevent the application of helmet or nasal cannula to patient's face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Inspiratory effort | 40 minutes
  The negative deflection in esophageal pressure during inspiration
Tidal volume | 40 minutes
  The tidal change in lung impedance, assessed by electrical impedance tomography

SECONDARY OUTCOMES:
Oxygenation | 40 minutes
  Ratio of PaO2 to FiO2
Tidal volume distribution | 40 minutes
  Distribution of tidal volume within the lung regions, assessed by electrical impedance tomography
Carbon dioxide | 40 minutes
  Blood carbon dioxide, measured with the arterial blood gas analysis
Respiratory rate | 40 minutes
  Respiratory rate/minute, assessed with the esophageal pressure
Dyspnea | 40 minutes
  Dyspnea assessed with the visual analog scale, 0-10 scale where the highest value corresponds to the highest degree of dyspnea
Comfort | 40 minutes
  Comfort assessed with the visual analog scale, 0-10 scale where the highest value corresponds to the highest degree of discomfort
Global impedance-derived End-expiratory lung volume | 40 minutes
  End-expiratory lung volume, measured with electrical impedance tomography
Regional impedance-derived End-expiratory lung volume | 40 minutes
  End-expiratory lung impedance in the four regions of the lungs (ventral, mid-ventral, mid-dorsal, dorsal), measured with electrical impedance tomography
Dynamic transpulmonary driving pressure | 40 minutes
  The tidal change in transpulmonary pressure
Global impedance-derived lung dynamic strain | 40 minutes
  Change in impedance due to tidal volume / end expiratory lung impedance, both measured with electrical impedance tomography
Regional impedance-derived lung dynamic strain | 40 minutes
  Change in impedance due to tidal volume / end expiratory lung impedance in the four regions of the lungs (ventral, mid-ventral, mid-dorsal, dorsal), measured with electrical impedance tomography
Respiratory system dynamic compliance | 40 minutes
  Ratio of the tidal change in lung impedance to dynamic transpulmonary driving pressure
Pendelluft | 40 minutes
  Occurrence of intra-tidal shift of gas within different lung regions at beginning of inspiration
Work of breathing | 40 minutes
  Esophageal pressure simplified pressure time product per minute

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS; Domenico L Grieco, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon a reasonable request

REFERENCES:
- [Derived] Menga LS, Delle Cese L, Rosa T, Cesarano M, Scarascia R, Michi T, Biasucci DG, Ruggiero E, Dell'Anna AM, Cutuli SL, Tanzarella ES, Pintaudi G, De Pascale G, Sandroni C, Maggiore SM, Grieco DL, Antonelli M. Respective Effects of Helmet Pressure Support, Continuous Positive Airway Pressure, and Nasal High-Flow in Hypoxemic Respiratory Failure: A Randomized Crossover Clinical Trial. Am J Respir Crit Care Med. 2023 May 15;207(10):1310-1323. doi: 10.1164/rccm.202204-0629OC. PMID 36378814